CLINICAL TRIAL: NCT05810298
Title: Effects of Pranayam (Voluntary Regulated Breathing) and Yogasana (Yoga Postures) on Posture, Pulmonary Parameters, Spine Flexibility, Body Awareness and Quality of Life Among Chronic Smokers
Brief Title: Effects of Yoga on Pulmonary Parameters, Posture, Body Awareness and Quality of Life Among Chronic Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CanerÖ
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Smoking
Keywords: Yoga; Pranayam; Breathing exercise; Asana; Smoking; Spine health; Spinal stretches
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers Group (Experimental): Education about smoking
  Asana practice (Only standing yoga poses with rhytmic breathing)
  Pranayam (Rhytmic regulated breathing)
  Interventions: Other: Asana Practice; Other: Pranayam Practice (Rhythmic regulated breathing); Behavioral: Smoking Education Program
- Control Group (Active Comparator): Asana practice (Only standing yoga poses with rhytmic breathing)
  Pranayam (Rhytmic regulated breathing)
  Interventions: Other: Asana Practice; Other: Pranayam Practice (Rhythmic regulated breathing)

INTERVENTIONS:
Other: Asana Practice — Yogasana training will be comprised of active movements when standing. Spine and limbs stretches eccentrically respecting the movement patterns of body without pushing limits. Transition in between poses will be synchronized with breathing pattern in zero resistance flow. The exercises will be done 2 days a week online under the supervision of physiotherapist. Total duration of standing poses training will last for 4 weeks.
Other: Pranayam Practice (Rhythmic regulated breathing) — Breathing exercises will be comprised of diaphragmatic breathing, holding the breath after inhaling deeply and exhaling passively or exhaling actively by contracting abdominal muscles and inhaling passively. The exercises will be done 2 days a week online under the supervision of physiotherapist. Total duration of breathing exercises will last for 4 weeks.
Behavioral: Smoking Education Program — The aim of the education is to increase awareness of subjects who are chronical smokers. The subject education will be performed at least once via face to face interview. Education topics will be covered basic information about harmful effects of habitual smoking and how to reduce the side effects of nicotine withdrawal.
  Arms: Smokers Group

SUMMARY:
The aim of this study is to examine the effects of practicing pranayam (voluntary regulated breathing) and yogasana (standing poses of yoga) with subject education on vital capacity, respiratory muscle strength, spinal flexibility, body awareness, quality of life and nicotine dependence of smokers and non-smokers.

DETAILED DESCRIPTION:
When initial assesments will be completed, volunteers will be assigned to one of two possible sequences by their nicotine dependency. Smokers group (SG) or control group (CG).

All volunteers will receive an exercise program with Asana and Pranayam practices with the duration of 4 weeks.

All subjects will be assessed in terms of functional capacity, pulmonary functions, thoracic spine range of motion, postural analysis, respiratory muscle strength, body awareness, quality of life and nicotine dependence at the baseline and at the end of the study. Data will be collected from all the subjects at baseline and at the end of the study (4 weeks) by the same physiotherapist who also will supervise the exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in research
* Young healthy subjects who were aged between 18-60 years with or without daily cigarette smoking habit

Exclusion Criteria:

* Allergic disorders or respiratory disorders
* History of a major surgery in the last 2 years
* Neurological diseases
* Cardiovascular diseases which are contraindicates exercise
* Fractures or orthopedic problems in upper or lower extremities
* Systemic rheumatical diseases(Rheumatoid Arthritis, Ankylosing Spondilitis etc.)

Systemic diseases and respiratory disorders will be ruled out in the selected subjects by taking their detailed history and by their thorough clinical examination by the researcher.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Fagerström Test for Nicotine Dependence | 4 weeks
  Nicotine dependence will be evaluated with this test
Thoracic Spine Range of Motion | 4 weeks
  Thoracic spinal elasticity will be evaluated with measuring rotational range of motion of T1-T2 spine using iPhone compass app. A strong and significant correlation was found between the Universel Goniometer and the Compass app by Furness et al. (2018), demonstrating good concurrent validity.
Pulmonary Function Tests | 4 weeks
  Medical International Research Spirodoc® Spiro spirometry will be used to evaluate pulmonary functions of volunteers.
Respiratory Muscle Strength | 4 weeks
  The Micro Medical Micro RPM respiratory pressure meter will be used to evaluate respiratory muscle strength.
New York Posture Rating Chart | 4 weeks
  Different parts of body will be screened by the physiotherapist and observation data will be used to evaluate volunteers posture.
World Health Organization Quality of Life Assesment (WHOQOL-BREF) | 4 weeks
  Turkish version of WHOQOL-BREF will be used in this study as given by WHO. This questionnaire will be used to provide numerical data on Quality of Life assesments of the volunteers.
Body Awareness Questionnaire(BAQ) | 4 weeks
  Body Awareness Questionnaire(BAQ) will be used to provide numerical data on subjects body awareness. A Turkish validity study of BAQ was performed by Karaca and it's valid as well as reliable.

CONTACTS AND LOCATIONS:
Locations (1):
- Fizyoram Physiotherapy Counseling Center, Istanbul, Turkey (Türkiye)